CLINICAL TRIAL: NCT00752856
Title: Nucleoside-Sparing Combination Therapy With Lopinavir/Ritonavir (LPV/r) + Raltegravir (RAL) vs. Efavirenz (EFV) + Tenofovir Disoproxil Fumarate + Emtricitabine (TDF/FTC) in Antiretroviral-Naïve Patients
Brief Title: Raltegravir + Lopinavir/Ritonavir Versus Efavirenz + Tenofovir + Emtricitabine in Treatment Naive Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: California HIV/AIDS Research Program (Other); Merck Sharp & Dohme LLC (Industry); Abbott (Industry)
Responsible Party: Principal Investigator, Sheldon Morris, Clinical Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCTG 589
Record Dates: First submitted 2008-09-13; First posted 2008-09-16 (Estimated); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: HIV Infections
Keywords: HIV treatment; Treatment-naive; Adult
MeSH Terms: conditions — HIV Infections | interventions — lopinavir-ritonavir drug combination; Raltegravir Potassium; Lopinavir; Ritonavir; Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; efavirenz; Tenofovir; Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 - Kaletra + Isentress taken twice daily (Experimental): Kaletra (lopinavir/ritonavir 400/100 mg) + Isentress (Raltegravir 400 mg) twice-daily
  Interventions: Drug: Kaletra + Isentress
- 2 - Atripla taken once daily (Active Comparator): Sustiva (EFV 600 mg), Viread (TDF 300 mg) and Emtriva (FTC 200 mg) taken as Atripla® once-daily
  Interventions: Drug: Atripla

INTERVENTIONS:
Drug: Kaletra + Isentress — kaletra 2 tabs twice a day + Raltegravir 1 tab twice a day
  Other Names: Lopinavir/ritonavir (LPV/r) + Raltegravir (RAL)
  Arms: 1 - Kaletra + Isentress taken twice daily
Drug: Atripla — Atripla 1 tab once a day
  Other Names: Efavirenz (EFV) + Tenofovir Disoproxil Fumarate + Emtricitabine (TDF/FTC)
  Arms: 2 - Atripla taken once daily

SUMMARY:
CCTG 589 is a randomized, open-label, pilot study comparing the efficacy, safety and tolerability of RAL plus LPV/r to EFV plus TDF/FTC in HIV-infected, treatment-naïve subjects. Subjects will be ineligible if they have any evidence of drug resistant virus in the past or at the time of screening (if never previously tested). Those who are found to be eligible will be randomized 1:1 to initiate either LPV/r (400/100 mg) plus RAL (400mg), both given twice-daily, or fixed dose combination of EFV (600 mg), TDF (300 mg) and FTC (200 mg) given as once-daily Atripla® for 48 weeks.

Hypotheses

1. The novel nucleoside-sparing combination of LPV/r + RAL will have a faster phase 1 viral decay rate compared to standard-of-care therapy with EFV/TDF/FTC in antiretroviral-naïve patients.

   1. Faster phase 1 viral decay dynamics will be associated with improved longer-term (week 48) viral suppression.
   2. Faster phase 1 viral decay dynamics will be associated with accelerated early (Day 0-14) clearance of cell-associated HIV DNA.
   3. Faster phase 1 viral decay dynamics will be associated with greater early (baseline to week 12) CD4+ T-cell recovery.
2. The LPV/r + RAL arm will have greater decreases in early (baseline to week 4) CD4/CD8 T-cell immune activation and apoptosis which will be associated with greater late (week 12 to week 48) CD4+ T-cell recovery.
3. Subjects treated with LPV/r + RAL arm will have smaller changes in total cholesterol and triglycerides from baseline than those receiving EFV/TDF/FTC.

DETAILED DESCRIPTION:
The purpose of this study is to determine how well a new anti-HIV drug combination (RAL plus LPV/r) taken twice a day decreases the amount of HIV found in participants' blood (viral load) compared to taking the once-a-day combination pill Atripla®. This study will also try to determine if the new combination has fewer side effects and is tolerated better than Atripla®. Another reason this study is being done is to see if this new drug combination helps participants' body's CD4 cells recover differently and will also look at how well participants' bodies absorbs these drugs and how safe these drugs are when given together.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection.
* Treatment naïve (defined as having never received any HIV antiretroviral agents in past).
* CD4+ T-cell count greater than or equal to 50 cells/mm3
* HIV viral load greater than or equal to 5,000 copies/mL
* Laboratory values obtained by screening laboratories within 30 days of entry:

  * Absolute neutrophil count (ANC) greater than 750/mm3.
  * Hemoglobin greater than 8.0 g/dL.
  * Platelet count greater than 50,000/mm3.
  * Calculated creatinine clearance (CrCl) > 60 mL/min as estimated by the Cockcroft-Gault equation:

    * For men, (140 - age in years) x (body weight in kg) ÷ (serum creatinine in mg/dL x 72) = CrCl (mL/min)
    * For women, multiply the result by 0.85 = CrCl (mL/min)
  * AST (SGOT), ALT (SGPT), and alkaline phosphatase less than 5 x ULN.
  * Total bilirubin less than 2.5 x ULN.
* Females of childbearing potential must have a negative serum pregnancy test at screening and agree to use a double-barrier method of contraception throughout the study period.
* Men and women age greater than or equal to 18 years.
* Ability to obtain prescription for HIV antiretroviral medications and to have required prescriptions filled prior to entry.
* Ability and willingness of subject to give written informed consent

Exclusion Criteria:

* Pregnancy or breast-feeding
* Serious illness requiring systemic treatment and/or hospitalization until subject either completes therapy or is clinically stable on therapy, in the opinion of the investigator, for at least 30 days prior to study entry (day 0).
* Acute therapy for serious infection or other serious medical illnesses (in the judgment of the site investigator) requiring systemic treatment and/or hospitalization within 14 days prior to study entry (day 0).
* Evidence of HIV seroconversion within 6 months prior to study entry.
* Evidence of any major HIV drug resistance-associated mutation on any genotype performed prior to study entry or at the time of screening.
* History of chronic hepatitis C (defined as HCV antibody positive and HCV RNA detectable).
* History of chronic active hepatitis B (defined as surface antigen positive and/or HBV DNA detectable).
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
* Use of any immunomodulator, HIV vaccine, or investigational therapy within 30 days of study entry.
* Use of human growth hormone within 30 days prior to study entry.
* Initiation of testosterone or anabolic steroids within 30 days prior to study entry. (Exception: Chronic replacement dosages in patient's with diagnosed hypogonadism is allowed).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2008-08-26 (Actual); Primary Completion 2011-05-05 (Actual); Study Completion 2014-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Haubrich, MD, Principal Investigator — California Collaborative Treatment Group (CCTG); Sheldon Morris, MD, Study Chair — UC San Diego AntiViral Research Center (AVRC)
Locations (6):
- United States (6):
  - Living Hope Clinical Foundation, Long Beach, California
  - University Southern California, Los Angeles, California
  - Univerisity California Irvine, Orange, California
  - Desert AIDS Project, Palm Springs, California
  - University California San Diego, San Diego, California
  - Harbor-UCLA, Torrance, California

REFERENCES:
- [Derived] Karris MY, Jain S, Bowman VQ, Rieg G, Goicoechea M, Dube MP, Kerkar S, Kemper C, Diamond C, Sun X, Daar ES, Haubrich RH, Morris S; California Collaborative Treatment Group (CCTG) 589 Study Team. Nucleoside-Sparing Regimens With Raltegravir and a Boosted Protease Inhibitor: An Unsettled Issue. J Acquir Immune Defic Syndr. 2016 Jun 1;72(2):e48-50. doi: 10.1097/QAI.0000000000000990. No abstract available. PMID 26977746

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1 - Kaletra + Isentress Taken Twice Daily | 2 - Atripla Taken Once Daily
Started | 26 | 25
Completed | 26 | 24
Not Completed | 0 | 1
Not completed — randomized but did not do viral kinetics | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 - Kaletra + Isentress Taken Twice Daily | 2 - Atripla Taken Once Daily | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 40 [30.3 to 47.5] | 43 [32.7 to 47.8] | 43 [31 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 25 | 24 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 21 | 22 | 43
  Black | 5 | 0 | 5
  Asian | 0 | 1 | 1
  Other | 0 | 2 | 2
  Hispanic | 12 | 14 | 26
  Non-Hispanic | 14 | 11 | 25

OUTCOME MEASURES:

1. Primary Outcome: To Compare the Phase 1 Viral Decay Rates Between LPV/r + RAL vs. EFV/TDF/FTC Treatment Combinations.
Description: Repeated HIV RNA measured at different time points (baseline, days 2, 7, 10, 14) will be treated as the outcome variable in a linear mixed-effects model. The primary fixed effects will include time, treatment group, treatment group-by-time interaction; random effects will include both intercept and slope allowing each subject to have individual baseline viral load and viral decay (rate of decrease in viral load following initiation of antiretroviral therapy). The treatment group-by- time interaction term in the model will indicate the difference in viral decay rates between the two treatment groups. Baseline covariate adjustment will be included if necessary.
Time Frame: Baseline, days 2, 7, 10, 14
Measure: Median (Inter-Quartile Range); unit: log(10)/day
Arm/Group | 1 - Kaletra + Isentress Taken Twice Daily | 2 - Atripla Taken Once Daily
Number analyzed (Participants) | 26 | 24
log(10)/day | 0.47 [0.42 to 0.52] | 0.55 [0.52 to 0.58]

2. Secondary Outcome: Viral Suppression Efficacy at 48 Weeks
Description: To determine the antiviral efficacy of LPV/r + RAL compared to EFV/TDF/FTC after 48 weeks of treatment by achieving undetectable viral load
Time Frame: 48 weeks
Measure: Number; unit: percentage of participants
Arm/Group | 1 - Kaletra + Isentress Taken Twice Daily | 2 - Atripla Taken Once Daily
Number analyzed (Participants) | 26 | 24
percentage of participants | 86 | 87.5

3. Secondary Outcome: Compare Early Activated CD4+ T-cell Recovery Rates From Baseline to Week 4.
Description: To compare early (baseline to Week 4) activated CD4+ T-cell recovery rates between treatment regimens.
Time Frame: Baseline to Week 4
Population: Participants who achieved viral suppression at week 24 and maintained it at week 48 were included in this analysis.
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | 1 - Kaletra + Isentress Taken Twice Daily | 2 - Atripla Taken Once Daily
Number analyzed (Participants) | 12 | 16
cells/mm^3 | -3.81 [-6.12 to -1.51] | -1.18 [-3.17 to 0.08]

4. Secondary Outcome: Compare Late Activated CD4+ T-cell Recovery Rates Between Treatment Regimens From Baseline to Week 48
Description: To compare late (baseline to Week 48) activated CD4+ T-cell recovery rates between treatment regimens.
Time Frame: 48 weeks
Population: Participants who achieved viral suppression at week 24 and maintained it at week 48 were included in this analysis.
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | 1 - Kaletra + Isentress Taken Twice Daily | 2 - Atripla Taken Once Daily
Number analyzed (Participants) | 12 | 16
cells/mm^3 | -2.24 [-5.83 to 1.36] | -5.65 [-8.76 to -2.54]

ADVERSE EVENTS:
Arm/Group | 1 - Kaletra + Isentress Taken Twice Daily | 2 - Atripla Taken Once Daily
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 13/26 | 15/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 - Kaletra + Isentress Taken Twice Daily (N=26) | 2 - Atripla Taken Once Daily (N=25)
Generalized Symptoms (General disorders) | 3 (4) | 4 (4)
GI Symptoms (Gastrointestinal disorders) | 13 (14) | 4 (4)
Pain, Aches & Muscle Discomfort (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5)
Any CNS Symptoms (Nervous system disorders) | 3 (3) | 14 (14)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2008-06-06): https://cdn.clinicaltrials.gov/large-docs/56/NCT00752856/Prot_SAP_000.pdf